CLINICAL TRIAL: NCT00839501
Title: Therapeutic Trial of Potassium and Acetazolamide in Andersen-Tawil Syndrome
Brief Title: Effect of Potassium and Acetazolamide on People With Andersen-Tawil Syndrome
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Unable to recruit sufficient number of participants
Sponsor: University of Rochester (Other)
Collaborators: Office of Rare Diseases (ORD) (NIH); Rare Diseases Clinical Research Network (Network); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Robert Griggs, MD, Professor of Neurology, Pediatrics, Pathology & Laboratory Medicine, and Center for Human Experimental Therapeutics, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: RDCRN 5305; U54NS059065 (NIH)
Record Dates: First submitted 2009-02-05; First posted 2009-02-09 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Andersen-Tawil Syndrome
MeSH Terms: conditions — Andersen Syndrome | interventions — Potassium; Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Participants will receive either potassium or placebo during six 3-week-long treatments, as randomly determined. Participants will then continue to receive potassium, if tolerated, and also either acetazolamide or placebo during another six 3-week-long treatments, as randomly determined.
  Interventions: Dietary Supplement: Potassium; Drug: Acetazolamide

INTERVENTIONS:
Dietary Supplement: Potassium — 40 mEq twice daily in pill form during the first 3-day inpatient visit, followed by 40 mEq twice daily in liquid form during the first 18-week treatment period, as is randomly scheduled, and continued during the second 18-week treatment period as long as there are no limiting side effects
Drug: Acetazolamide — 250 mg twice daily, orally, during the second 3-day inpatient visit and during the second 18-week treatment period, as is randomly scheduled

SUMMARY:
Andersen-Tawil Syndrome (ATS) is a rare genetic disorder that causes episodes of muscle weakness, potentially life-threatening changes in heart rhythm, and skeletal developmental abnormalities. The cause of some ATS cases remains unknown, and no specific treatments have been established. The purpose of this study is to determine whether potassium supplements and/or the medication acetazolamide affect the duration of muscle weakness and heart rhythm abnormalities in people with ATS.

DETAILED DESCRIPTION:
ATS is an ion channel disorder that causes episodes of muscle weakness and potentially life-threatening heart arrhythmias. The majority of ATS cases are caused by a mutation in the KCNJ2 gene, which is linked to potassium channels in the heart, brain, and skeletal muscle; other cases are presumed to be caused by an as yet undetermined gene lesion. To date, the treatment for ATS has been largely anecdotal, and no treatments have been formally assessed in a controlled clinical trial. This study will determine whether potassium supplements and/or acetazolamide, which is a diuretic medication, affect the duration of muscle weakness and heart rhythm abnormalities in people with ATS.

Participation in this study will last about 11 months. Participants will first attend a 3-day inpatient visit that will include a medical history, physical examination, blood work, heart rhythm testing by an electrocardiogram (ECG) and Holter monitor, strength testing, a health questionnaire, and daily potassium supplementation. Participants will also track the number and length of weakness episodes that they experience while in the hospital. On the last day of the inpatient visit, participants will be provided with multiple bottles containing either potassium or placebo. Participants will then return home for an 18-week treatment period that will consist of six 3-week-long treatments of either potassium or placebo, with the treatment schedule being randomly determined. Upon completing the first 18-week treatment period, participants will attend a second 3-day inpatient visit that will include the same tests and procedures as the first. The only difference will be that participants will receive acetazolamide along with potassium. This will be followed by a second 18-week treatment period that will consist of six 3-week-long treatments of either acetazolamide or placebo. At the end of the second treatment period, participants will fill out another health questionnaire. Throughout both 18-week treatment periods, participants will phone in daily to track any muscle or heart problems. They will also provide blood samples on a weekly basis. At Weeks 2, 5, 8, 11, 14, and 17 of both treatment periods, participants will wear a Holter monitor for 24 hours and then mail it in. A final outpatient visit will occur 8 weeks after the end of the second treatment period and will include heart rhythm testing, muscle strength testing, and blood work.

ELIGIBILITY:
Inclusion Criteria:

* Clinically confirmed diagnosis of Andersen-Tawil Syndrome, as defined by at least two of the following three features:

  1. Neuromuscular Feature

     * Presence of clear-cut episodes of transient muscle weakness with or without a fixed deficit that is typical with rest after exertion or prolonged rest, OR
     * An atypical history with specific exam findings (absent reflexes with normal sensation ictally), OR
     * Unexplained intraictal hypokalemia, OR
     * An abnormal nerve conduction exercise test
  2. Cardiac Feature

     * Prolonged QTc interval on 12-lead electrocardiogram (ECG), according to standard criteria, AND/OR
     * Ventricular ectopy, including uniform or multifocal PVCs, polymorphic VT, or bidirectional VT
  3. Physical Feature (at least two of the below five features)

     * Low set ears
     * Hypertelorism
     * Small mandible
     * Clinodactyly
     * Syndactyly
     * Micromelia of hands or feet

-OR-

* One of the three above criteria, with at leat one other family member meeting two criteria

-OR-

* Not meeting clinical criteria but possessing the KCNJ2 mutation
* An average frequency of at least one neuromuscular symptom (attack of weakness) per week

Exclusion Criteria:

* Sulfa allergy
* Renal impairment, as defined by serum creatine greater than 1.5 mg/dl
* History of renal calculi
* Cardiac disease or other disease that would make potassium supplementation or acetazolamide treatment inadvisable
* Diabetes mellitus
* Currently taking quinidine
* Pregnant

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-12; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Sum of the attack durations across the entire treatment period, reported by the participants via interactive voice response (IVR) | Measured over two 18-week treatments periods

CONTACTS AND LOCATIONS:
Overall Officials: Paul Twydell, DO, Principal Investigator — University of Rochester School of Medicine & Dentistry
Locations (1):
- University of Rochester School of Medicine, Rochester, New York, United States